CLINICAL TRIAL: NCT07319468
Title: Effect of Intra Dialytic Aerobic Exercises Versus Active Free Exercises on Cognitive Function and Functional Capacity in Hemodialytic Patients
Brief Title: Effect of Exercises on Hemodialysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Faten Mahmoud, Consultant of Physical Therapy, Chest Hospital, Damanhour, Elbeheira, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NO:P.T.R.EC/012/004902
Record Dates: First submitted 2025-12-09; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Hemodialytic Patients
Keywords: Aerobic Exercise; Chronic kidney disease; Hemodialysis; Functional Capacity
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic exercise (Experimental): (23) patients who received aerobic exercise in form of (foot pedal exerciser) for 20 Minutes for each session, 3 sessions per week, for 8 weeks.
  Interventions: Device: Aerobic exercises
- Active free range of motion exercise (Experimental): (23) patients who received active free range of motion exercise (open kinetic chain active free range of motion) for 20 minutes for each session, 3 sessions per week, for 8 weeks.
  Interventions: Other: Open kinetic chain active free range of motion
- control group (Other): (23) patients who will receive standard medical treatment for end-stage renal disease, including regular hemodialysis sessions and pharmacological management (e.g., Epoetin alfa and phosphate binders) as prescribed by their nephrologist, without participating in the physical therapy exercise program.
  Interventions: Other: No intervention

INTERVENTIONS:
Device: Aerobic exercises — Foot pedal exerciser:
  * Simple horizontal foot pedal exerciser used during hemodialysis sessions.
  * Dual pedals with non-slip straps for foot stability.
  * Manual resistance adjustment via a single control knob (non-electric).
  * Provides gradual increase in workload intensity.
  * Compact and light weight design suitable for use while lying on the dialysis bed.
  * Enables controlled, low-impact circular movement of the feet.
  * Aims to improve circulation and strengthen lower limb muscles without requiring active sitting.
  * Approximate device dimensions: 50 cm (length) x 40 cm (width) x 23 cm (height).
  * Maximum recommended user weight: 70 kg.
  Arms: Aerobic exercise
Other: Open kinetic chain active free range of motion — Participants completed the 30-min aerobic exercise sessions during the first 2 hrs. of each dialysis session, 3 times per week for 8 weeks, using a simulated bike riding. Patients will perform active free exercise for upper limb (the arm that hasn't shunt) and lower limbs. Each exercise session consisted of three phases: warm up, conditioning, and cool down.
  Arms: Active free range of motion exercise
Other: No intervention — the control group will receive only the standard medical care provided by dialysis center without any physical therapy intervention
  Arms: control group

SUMMARY:
o Sixty-nine adult patients from both sexes. They were suffering from ESRD on maintenance hemodialysis, their age ranged from50-60 years old were selected from hemodialysis unit at Itay El Baroud central hospital. They were referred by the physician.

DETAILED DESCRIPTION:
Ⅰ-Subjects:

o Sixty-nine adult patients from both sexes. They were suffering from ESRD on maintenance hemodialysis, their age ranged from50-60 years old were selected from hemodialysis unit at Itay El Baroud central hospital. They were referred by the physician.

Study group (A): the study group consisted of (23) patients who received aerobic exercise in form of (foot pedal exerciser) for 20 Minutes for each session, 3 sessions per week, for 8 weeks plus maintain on their medical treatment and hemodialysis.

Study group (B): the study group consisted of (23) who received active free range of motion exercise (open kinetic chain active free range of motion) for 20 minutes for each session, 3 sessions per week, for 8 weeks plus maintain on their medical treatment and hemodialysis.

Control group (C): the control group consisted of (23) patients who were maintained on their medical treatment and hemodialysis.

II- Instrumentation 6-Minutes walk test: The 6-min walk test (6MWT) is frequently used to measure physical function in transplanted patients.

* Fatigue Questionnaire (Fatigue Severity Scale) it was used to assess the level of fatigue.
* Laboratory investigation: urea and creatinine are commonly used to monitor the effects of exercise on urea clearance and kidney function improvement in transplant patients.
* The Mini-Cog test: is a quick, simple, and effective screening tool for early cognitive impairment in hemodialysis patients, making it ideal for busy clinical settings.

B-Therapeutic Equipment:

Foot pedal exerciser (fig.9):

* Simple horizontal foot pedal exerciser used during hemodialysis sessions.
* Dual pedals with non-slip straps for foot stability.
* Manual resistance adjustment via a single control knob (non-electric).
* Provides gradual increase in workload intensity.
* Compact and light weight design suitable for use while lying on the dialysis bed.
* Enables controlled, low-impact circular movement of the feet.
* Aims to improve circulation and strengthen lower limb muscles without requiring active sitting.
* Approximate device dimensions: 50 cm (length) x 40 cm (width) x 23 cm (height).
* Maximum recommended user weight: 70 kg. Participants completed the 30-min aerobic exercise sessions during the first 2 hrs. of each dialysis session, 3 times per week for 8 weeks, using a simulated bike riding. Patients will perform active free exercise for upper limb (the arm that hasn't shunt) and lower limbs. Each exercise session consisted of three phases: warm up, conditioning, and cool down.

ELIGIBILITY:
Inclusion Criteria:

All patients were included according to the following criteria:

1. Age between 50-60years.
2. The patients had been on hemodialysis for at least 3 months with three sessions per week for 3-4hr per session.
3. The patients were diagnosed with end stage renal failure (stage5 CKD) on maintenance regular HD (three sessions/week (on alternate days), for four hours/session) for more than three months. (Receiving HD through uncomplicated arm arteriovenous (A-V) fistula
4. Under medical control
5. Both men and women were enrolled
6. Body math index ranged from 18,5- 24.9 kg/m²

Exclusion Criteria:

Patients who experienced or had one or more of the following were excluded from the study:

1. Patients with resting systolic blood pressure >200 mmHg and/or diastolic blood pressure >120 mmHg.
2. patients with neurological problems (e.g. stroke, head injury)
3. patients with musculoskeletal problems (e.g. sever osteoarthritis or difficulties in ambulation)
4. Patients with uncontrolled pulmonary disease. (e.g. exaggerated chronic obstructive pulmonary disease, acute asthma)
5. Patients with mental health problems and cognitive impairment due to inability to teach them how to make respiratory training.
6. Any patient who missed more than two weeks of the program or want to terminate the program.
7. Severe obesity (BMI >35)
8. Presence of malignant disease.
9. Patients with unstable angina, uncontrolled cardiac arrhythmia, decompensated heart failure, acute pericarditis or myocarditis.
10. The patients had hearing impairment or mental disorders.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue Questionnaire (Fatigue Severity Scale) | 8 weeks
  The Fatigue Severity Scale it used to assess the level of fatigue. The Fatigue Severity Scale scores range from 9 to 36 where higher scores indicate worse fatigue and lower scores indicate improvement in fatigue.
6-Minutes walk test | 8 weeks
  The 6-min walk test (6MWT) is frequently used to measure physical function in transplanted patients

SECONDARY OUTCOMES:
Laboratory investigation (Urea analysis) | 8 weeks
  Urea analysis is commonly used to monitor the effects of exercise on urea clearance and kidney function
The Mini-Cog test | 8 weeks
  The Mini-Cog test is a quick, simple, and effective screening tool for early cognitive impairment in hemodialysis patients, making it ideal for busy clinical settings. The Mini-Cog Test scores range from 0 to 5, where higher scores indicate better cognitive performance, and lower scores suggest potential cognitive impairment.
Laboratory investigation (creatinine analysis) | 8 weeks
  creatinine analysis is used to be monitor the effects of exercise on creatinine clearance and kidney function

CONTACTS AND LOCATIONS:
Overall Officials: Research Ethical Committee Cairo University, Principal Investigator — Cairo University